CLINICAL TRIAL: NCT02336412
Title: The Use of Short Message Service (SMS) as a Reminder for Continuation of Treatment With Secondary Preventative Medications After Stroke or TIA
Brief Title: Short Message Service (SMS) Reminders for Stroke Secondary Preventative Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GN14NE625
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Stroke; Ischemic Attack, Transient
Keywords: Medication adherence
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS reminder (Experimental): Daily SMS medication reminder
  Interventions: Other: SMS reminder
- No SMS reminder (No Intervention): No daily SMS medication reminder

INTERVENTIONS:
Other: SMS reminder — Daily SMS medication reminder
  Arms: SMS reminder

SUMMARY:
Secondary preventative medications are prescribed to reduce the risk of recurrent stroke following ischaemic stroke. However, continuation rates can be as low as 50% and are likely to be multifactorial. One factor will be patients forgetting to take the medication or a reduced appreciation of the importance of the medication as the time from the stroke passes. Numerous approaches to improve persistence to secondary preventative medications have been tried. One simple approach is use of mobile phone text messages as a reminder for patients to take their medications. In this study, we will introduce an educational and motivational strategy to inform patients about their medications and explore whether a reminder intervention, using Short Message Service (SMS), improves adherence to antiplatelet drugs, antihypertensive medications and lipid lowering drugs. We will also explore whether this improves blood pressure and cholesterol levels in the first 3 months after stroke.

DETAILED DESCRIPTION:
We aim to recruit adult patients diagnosed with stroke or transient ischaemic attack (TIA) who were prescribed secondary preventative medication and are living in the community. They will be provided with a patient information sheet (PIS) with details on the study and will be contacted later to ask if they wish to take part. If so, an arrangement will be made for them to attend a clinic review where they will sign the consent form. Immediately then participants who consent will be randomized into control (will receive education and motivation interviews but not text messages to remind them) or intervention (will receive education and motivation interviews and will be sent a daily text message to remind them of taking their medication). Baseline assessment will include medical history and medications prescribed. They will be given detailed information on their specific prescribed medication and will be handed booklets with relevant information. They will be asked to answer a medication adherence questionnaire and will be given a medication diary to fill in at home. All participants will receive ambulatory blood pressure monitoring.

Cholesterol measurement will be made using a finger prick monitor. Participants in the intervention group will be informed that they will receive a daily text message in the morning to remind them about their medications.

Follow-up visits will take place after 1 and 3 months in which the same checks will be carried out as at the baseline visit. At 1 month, the cholesterol level and ambulatory blood pressure level will be repeated. Participants will be encouraged to ask if they have any concerns regarding their medications. At the end of the second visit, participants will be asked if they are satisfied with the care they received during the visits as a quality assessment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stroke or TIA
* treated with any combination of anti-platelet, antihypertensive, and/or lipid-modifying drugs; at least one of which started over the past month
* living in the community

Exclusion Criteria:

* severe disability (modified Rankin Scale (mRS) ≥ 4)
* patients unable to consent
* patients with no facility to be reminded by SMS or voicemail message

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Adherence rate to stroke secondary preventative medication | 3 months
  Morisky Medication Adherence Scale (MMAS) - 8 items

SECONDARY OUTCOMES:
Effect of medication adherence on clinical outcomes | 3 months
  Number of participants reaching target blood pressure level
Effect of medication adherence on clinical outcomes | 3 months
  Number of participants reaching target cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dawson, BSc MBChB MD, Study Director — University of Glasgow
Locations (1):
- Western Infirmary, NHS Greater Glasgow and Clyde, Glasgow, United Kingdom